CLINICAL TRIAL: NCT02258048
Title: The Use of Transient Elastography to Predict Clinical Decompensation in Patients With Early Cirrhosis
Status: Withdrawn | Type: Observational
Why Stopped: Samuel Sigal no longer with NYU
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 10-02236
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Cirrhosis
Keywords: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cirrhosis

SUMMARY:
This is a prospective study designed to examine the role of transient elastography as a predictor of clinical decompensation in patients with early cirrhosis. The study objective is to determine if changes in measurements of liver stiffness with transient elastography can identify patients that will have a more rapid progression of cirrhosis and the development of clinical decompensation. The target population is patients with early stage, well-compensated cirrhosis.

Participants of this study will be asked to complete the following procedures: read and sign the informed consent, medical records review (complete medical history, physical examination, laboratory evaluation, endoscopic findings, radiographic findings), undergo transient elastography to measure liver stiffness every three months until the development of clinical decompensation (ascites, variceal bleeding, hepatorenal syndrome, overt hepatic encephalopathy) for up to 2 years.

DETAILED DESCRIPTION:
This is a prospective study designed to examine the role of transient elastography as a predictor of clinical decompensation in patients with early cirrhosis. The study objective is to determine if changes in measurements of liver stiffness with transient elastography can identify patients that will have a more rapid progression of cirrhosis and the development of clinical decompensation. The target population is patients with early stage, well-compensated cirrhosis.

This study will attempt to determine if serial measurements of liver stiffness with transient elastography in patients with early cirrhosis can identify patients at risk of morbidity or mortality associated with hepatic decompensation.

For the Screening Visit, the following procedures will be performed:

1. Patient will read and sign informed consent. Subjects will be given sufficient time to consider, ask questions, and sign the consent forms.
2. Patient will be assigned a subject number
3. Patient will be asked to provide demographic information
4. Patient will be asked to provide a complete medical history and laboratory evaluation
5. Physical examination including blood pressure, heart rate, height, and weight.
6. The following assessments will also be performed:

   * Calculation of modified Child Pugh Score: Using the following biochemical variables: Serum Albumin, Total Bilirubin, Serum Creatinine, and INR.
   * MELD Score: Based on a continuous function of Bilirubin, INR, and Creatinine, which uses a continuous variable ranging from 6-40.
7. 30cc of blood will be obtained, and serum frozen at -80C (freezer located in Dr. Sigal's office) for up to 5 years. The blood will only be accessible to Dr. Sigal and his research team. This blood may be analysed for known markers of liver disease, markers that may be discovered in the future, and/or to identify new markers of liver disease.

For the Follow-Up Visits the following procedures will be performed every 3 months for up to 2 years:

1. An interim medical history will be obtained, with particular attention to the development of clinical decompensation (ascites, variceal bleeding hepatorenal syndrome, overt hepatic encephalopathy).
2. Physical examination.
3. Measurement of liver stiffness using hepatic elastography.
4. 30cc of blood will be obtained, and serum frozen for future analyses as above.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients with histologic or radiographic evidence of cirrhosis will be screened for participation in the study.
* Able to provide informed consent
* MELD score <10
* No history of ascites, variceal bleeding, hepatorenal syndrome, overt hepatic encephalopathy.

Exclusion Criteria:

* History of variceal bleeding, ascites, hepatorenal syndrome, or overt hepatic encephalopathy
* Inability to provide informed consent
* Body mass index (BMI)>35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients with histologic or radiographic evidence of cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Liver Stiffness | 2 years
  Liver stiffness will be measured using hepatic elastography.

SECONDARY OUTCOMES:
Evidence of Portal Hypertension | 2 years
  Presence of significant portal hypertension will be determined by the presence of ascites or thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, M.D., Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States